CLINICAL TRIAL: NCT05930704
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-dose, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SHR-2017 Injection Administered Subcutaneously to Postmenopausal Women
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SHR-2017 Injection in Postmenopausal Women
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR-2017-101
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-2017 injection (Experimental)
  Interventions: Drug: SHR-2017 injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-2017 injection — Randomized participants of multiple dose cohorts will receive a single subcutaneous dose of SHR-2017 injection.
  Arms: SHR-2017 injection
Drug: Placebo — Randomized participants will receive a single SC injection dose of matching placebo.
  Arms: Placebo

SUMMARY:
The primary objective was to evaluate the safety and tolerability of SHR-2017 after a single subcutaneous (SC) injection in postmenopausal women

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women ages ≥ 50 years.
2. Body weight≥45 kg, body mass index (BMI) of 18.0 to 29.0 kg/m2 (inclusive).
3. Understand in detail the content, procedure and possible adverse effects of the trial, and voluntarily sign the written informed consent form (ICF).

Exclusion Criteria:

1. History of malignancy.
2. Menopause due to simple hysterectomy.
3. Subjects with poor blood pressure control.
4. Subjects with positive tests for infectious diseases.
5. Have a history of diseases related to bone metabolism.
6. Use of drugs that may affect bone metabolism before administration.
7. Have a history of alcoholism, medical abuse, or drug use, or have a positive alcohol breath test or drug abuse screening.
8. Female who are pregnant or breastfeeding.
9. Unable to tolerate venipunctures or have a history of fainting needles and blood.
10. Other reasons that the investigator consider it inappropriate to participate in the trial.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-04-12 (Estimated); Study Completion 2025-04-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | From day 1 up to 9 months

SECONDARY OUTCOMES:
Maximum observed concentration of SHR-2017 (Cmax) | Day 1 pre-dose up to Day 253
Area under the serum concentration time curve from time 0 to time of last quantifiable serum concentration (AUC0-t) of SHR-2017 | Day 1 pre-dose up to Day 253
Time to maximum observed concentration (Tmax) of SHR-2017 | Day 1 pre-dose up to Day 253
Percent change from baseline in Urinary N-Telopeptide Corrected for Urine Creatinine (uNTx/Cr) | Baseline up to Day 253
Percent change from baseline in serum Type I Collagen Carboxy-terminal Peptide (CTX) | Baseline up to Day 253
Percent change from baseline in Intact Parathyroid Hormone (iPTH) | Baseline up to Day 253
Percent change from baseline in Bone-Specific Alkaline Phosphatase (BALP) | Baseline up to Day 253
Number of subjects who developed SHR-2017 antidrug antibodies (ADA) | Baseline up to Day 253

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shangdong, China

IPD SHARING:
Plan to Share IPD: Undecided